CLINICAL TRIAL: NCT01695200
Title: The Role of Omega-3 Fatty Acids in the Management of Singaporean Children With Autism Spectrum Disorders
Brief Title: Omega-3 Fatty Acids in Autism Spectrum Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Healthcare Group, Singapore (Other Government)
Responsible Party: Principal Investigator, Dr. Sung Min, Senior Consultant, National Healthcare Group, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSRB: 2011/00028
Record Dates: First submitted 2012-09-21; First posted 2012-09-27 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omega-3 Fatty Acids (Experimental): 15ml omega-3 liquid form, twice a day for 12 weeks (Total daily dosage:840mg DHA and 192mg EPA)
  Interventions: Dietary Supplement: Omega-3 fatty acids

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acids

SUMMARY:
This is a 12-week open label trial to evaluate whether omega-3 fatty acids is effective in reducing the severity of autism and its comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 5 and 18 years old
* Diagnosed to have Autism, Asperger Syndrome, or PDDNOS by the DSM-IV criteria; met the Autism or Spectrum classification for Autism Diagnostic Interview - Revised (ADI-R) and Autism Diagnostic Observation Schedule (ADOS)
* Written parental consent for participation
* Those not on current standard-of-care treatments for ASD

Exclusion Criteria:

* Below 5 and above 18 years old
* No formal diagnosis of Autism, Asperger Syndrome or PDD-NOS
* Without written parental consent for participation
* Those with brain pathology such as serious head injury, epilepsy, etc.
* Those on current standard-of-care treatment for ASD
* Those with psychotic symptoms, self-injurious behaviours and/or suicidal tendency, and other history of clinically significant medical conditions screened by the attending doctor to have increase the risk associated with study participation
* Those on other types of medication or supplements or with change in dose

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in parent rated Social Responsiveness Scale (SRS) scores during treatment | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in parent rated Child Behavior Checklist (CBCL) scores during treatment | 12 weeks
Change from baseline in teacher rated Teacher Report (TRF) scores during treatment | 12 weeks
Change from baseline in teacher rated Social Responsiveness Scale (SRS) scores during treatment | 12 weeks
Change from baseline in clinician rated Clinical Global Impression (Severity and Improvements) scores during treatment | 12 weeks
Change from baseline in clinician rated Global Assessment of Functioning (GAF) scores during treatment | 12 weeks
Children's Yale-Brown Obsessive Compulsive Scale modified for Pervasive Developmental Disorders (CYBOCS-PDD) | 12 weeks

OTHER OUTCOMES:
Assessment of plasma fatty acid composition, measurements of DHA and EPA (components of omega-3), and total phospholipid count | 12 weeks
Assessment of dietary intake and nutritional intake of the child | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Min Sung, MBBS, MMed, Principal Investigator — National Healthcare Group, Singapore
Locations (1):
- Institute of Mental Health, Singapore, Singapore